CLINICAL TRIAL: NCT00566267
Title: A Randomized, Double-Blinded Study of Simvastatin 20 mg/Day Versus Vytorin 10/20 in Subjects With Lipid Profiles Not Meeting Current NCEP Guidelines, Following a Low-Carbohydrate Diet
Acronym: LOCUST
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Frederick F. Samaha, M.D.
Organization: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 00887; MIRB Number: 00887; PROM # 0025
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2007-12-03 (Estimated); Status verified 2007-11

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Simvastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Experimental): Low carb diet plus simvastatin 20 mg/ezetimibe 10 mg
  Interventions: Drug: simvastatin 20 mg/ezetimibe

INTERVENTIONS:
Drug: simvastatin 20 mg/ezetimibe — see protocol
  Other Names: Low carb diet plus simvastatin 20 mg

SUMMARY:
People who follow a low-carbohydrate diet typically experience a decrease in triglycerides and increase in HDL-C level, but fail to lower their LDL cholesterol (LDL-C). Such patients may require lipid-lowering therapy. Statins may not be the most effective strategy for patients on this diet, since they typically consume a greater amount of saturated fat and cholesterol. Absorbed cholesterol may contribute more to their circulating plasma LDL-C. We hypothesize that patients following a low carbohydrate diet would experience a significantly greater decrease in LDL-C by taking ezetimibe 10 mg, a drug that blocks cholesterol uptake in the intestine, in addition to simvastatin 20 mg, when compared to taking simvastatin 20 mg alone.

ELIGIBILITY:
Inclusion Criteria:

* Moderately obese with hyperlipidemia

Exclusion Criteria:

* Recent unstable heart or lung condition
* Current use of other lipid modifying drugs
* Hepatic disease
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-04; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | 8 weeks of treatment

SECONDARY OUTCOMES:
Other lipid measures | 8 weeks of treatment
Safety and tolerability | 8 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frederick F Samaha, M.D., Principal Investigator — Philadelphia VAMC

REFERENCES:
- [Derived] Chirinos JA, Williams MM, Bregman DB, Ashfaq H, Khayyam U, Iqbal N. Efficacy of cholesterol uptake inhibition added to statin therapy among subjects following a low-carbohydrate diet: a randomized controlled trial. Am Heart J. 2010 May;159(5):918.e1-6. doi: 10.1016/j.ahj.2010.02.010. PMID 20435205